CLINICAL TRIAL: NCT02731781
Title: Trauma Infant Neurological Score (TINS) as a Prognostic Factor and Guideline for CT Scan in Infants 24 Months Old or Less
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Laniado Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 0130-15-LND
Record Dates: First submitted 2016-04-03; First posted 2016-04-08 (Estimated); Last update posted 2016-04-08 (Estimated); Status verified 2016-04

CONDITIONS: TO FIND THE CORRELATION BETWEEN TINS SCORE OUTCOME
Keywords: OUTCOME; PROGNOSIS; PEDIATRIC HEAd injury; CT SCAN

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: NONE . OBSERVATIONAL — OBSEVATION AND FOLLOW UP

SUMMARY:
Traumatic brain injury (TBI) is the major cause of disability and death among the younger population. In the Pediatric population Head trauma may be responsible for primary and secondary brain damage. Primary brain injury results from a direct mechanical damage at the time of injury, whereas secondary injury is caused by further cellular damage that develops hours or days post injury. Intracranial Injury in Infants (III) may be hard to diagnose in the abcence of neurological deficit or early deterioration. On the other hand, symptoms such as vomiting and restlessness may be present even in the case of minor head injury, and unnesessary scaning (CT) may be performed in many centers just because clinical judgment is problematic in this particular age. Some intracranial injuries may be imminent, such as evolving Epidural hematoma (EDH) in infants, and early diagnosis may be lifesaving and leading to excellent outcome. In adults, GCS has been accepted as the most usuful tool for emergency evaluation of head injured patients. In children, several scores were introduced, including the Children's Coma Score (CCS), however they have been found problematic to use in the very young population, since accurate evaluation of communication in CCS is hard, and there is insufficient relevant parameters uncorporated into the score that may have significant importance in this particular age group. In TINS (Trauma Infant Neurological Score) we characterized the clinical parameters and the mechanism of trauma in a simplified method. As previously published, this score has been used by us and by other groups, in retrospective studies. Still, in the lack of prospective studies using TINS, there are no optimal guidelines to perform computed tomography (CT) in this unique population, and TINS has not prospectively been challenged as a predictor tool for outcome. In this prospective study we will approach these issues.

DETAILED DESCRIPTION:
Methods:

200 infants (<2 years old) will be enrolled into the study. Clinical data will be gathered from the emergency room file, and in case of admission from the discharge letter and the clinical file. Based on the current protocols of treatment and diagnosis of children with head injury, CT will be performed according to the current axisting protocols. No intervention, imaging, or treatment will be administered different from the current protocol used in the hospital, according to the existing guidelines. Both TINS and Children's Glasgow Coma Scale (CCS) score was applied, based on the clinical data obtained from the files. If imaging is peformed data will be recoreded. As all children with head trauma are invited routinely to follow-up clinic within the 1st year after injury, this data will be recoreded as well.

As there is no violation of current treatment protocols, or any additional exams or interventions due to the study - and since the data is obtained from the files, informed concent will not be necessary.

The data will be coded by the treating doctors into a database that will be coded in a manner that identification of the child is not possible by the statisticians or by people who are not involved in treatment and follw up.

The database used will be a "filemaker pro" data base, with concequent numbering of the infant enrolled.

The difficulty in clinical assessment and early diagnosis of infants using different versions of the CCS, is well known as reported previously. [12-18] In our series, about half of the patients were brought in unconscious, whereas two infants had CCS scores of 15 on arrival and were neurologically intact .

In patients with no neurologic deficit and full alertness, a conservative approach may be chosen. Conservative treatment of acute epidural or subdural hematomas is rare. [20] This is usually suggested in patients with a small EDH (less than 1 cm thick and less than 3 cm in length in the anteroposterior plane on CT). If the patient is symptomatic, however (even severe headache present without any focal neurologic deficit), and the EDH is larger than 1 cm thick, surgery is the treatment of choice. In infants, symptoms are not always clear unless irritability or somnolence is observed. Objective signs rather than symptoms thus may be more helpful. If conservative treatment is chosen for an infant on admission, very close observation in an intensive care unit is mandatory. Also, in such cases, because of the lack of language communication and underestimation of symptoms, repeat CT is advised within 12 to 24 hours, even if no neurologic deterioration appears. As described above, one of the infants, a 7-month-old girl, was admitted with bilateral EDH. Conservative treatment was undertaken, with close observation; however, there was no neurologic deterioration during the subsequent 13 hours. On the next morning, repeat CT was performed, which clearly showed enlargement of the EDH on the left. The infant was then taken to the operating room, and bilateral craniotomy was performed. She was discharged within a few days in excellent condition with no neurologic deficit. In this rare example, the hematoma grew on CT without clinical deterioration, and surgery was indicated because the hematoma enlarged. Probably, the child would have deteriorated at a certain point because of the enlarging hematoma, but this was avoided by the routine repeat CT indicated in cases of attempted conservative treatment.

General Symptoms Transient loss of consciousness is not always clear in this age group, and lack of symptoms and signs in a fully awake baby may be confusing. [3-6,12] In our series, vomiting and loss of consciousness were very common. Also, most of the infants had significant subgaleal hematomas. In fact, in some infants, these were the only positive parameters for which CT was performed by the neurosurgeon, considering the young age of the patients.

CCS Score Looking at prognosis and CCS score on admission, one may be surprised. Of the five infants who arrived unconscious, three left the hospital neurologically intact. As was reported in previous series, a low CCS score in infants does not necessarily indicate a poor prognosis or gross neurologic deficits on discharge. [12,13] On the other hand, early diagnosis of EDH in infants admitted in good neurologic condition with a history of minor head injury is difficult. Neither good condition nor minor trauma can rule out an intracranial emergency. [13,17]

Mechanism of Injury In our series, most of the patients fell from less than 1 m, and even when they arrived in good neurologic condition, surgical EDH was found on CT. When mechanism of injury was a fall from more than 1 m, clinical presentation was much worse, with lateralizing signs, loss of consciousness, and a high rate of posterior fossa hematomas. This shows how vulnerable infants may be compared with older children even after minor head injury. A relatively high rate of posterior fossa EDH was found in our series compared with previous reports. [2-5,15]

Lag Time An interesting observation was the lag time we found (up to 48 hours) in some infants between the time of injury and admission to the ER. This was common with younger infants when parents at first underestimated the apparently minor head injury (fall from less than 1 m). These infants were eventually brought to the ER, however, because of some deterioration or unusual behavior. Another lag time was observed between admission to the ER and operation. This lag time was probably attributable to the good neurologic condition of some infants on admission. Less than half of the infants were operated on immediately on arrival or within 1 hour of presentation to the ER. This may suggest a rather subacute presentation of EDH in infants compared with children and adults. It can be explained either by better compliance of the infant cranium and brain, which delayed the appearance of severe symptoms, or by underestimation of the injury by the parents and the doctor as well.

Scoring Method for Infants Several Children's Coma Scales have been suggested in the past [1,7-11,21] to improve the neurologic evaluation of children compared with adults. When applied to infants, however, these scoring methods may be disappointing. An anatomic difference of skull size and flexibility, as well as the opened sutures and fontanels in infants, make the dynamics of the intracranial compartment different from that of older children. They may be more fragile but also more compliant. The pathophysiology of the evolving intracranial bleeding, in our case the EDH, thus may be different in both the form and the timing of clinical symptoms. [13,22-24]

One reason why application of CCS may be inaccurate and problematic for infants is that most suggested Children's Coma Scales include parameters that are difficult to interpret and score. Examples are infants' interaction with the examiner, restlessness or consolability, and the difficult evaluation of sound and cry. The problem is greater than in older children because infants' psychomotor development is variable (each infant has a different speed and level) and verbal communication is incomplete-considerations that may influence the CCS applied. We think that in this age group, therefore, objective parameters, which are clear and evident to any examiner, should be used.

The New Trauma Infant Neurologic Score IN 1999 new approach and scoring system was proposed and reported by Beni Adani et all (Ref 25), that is not necessarily a tailored or revised Glasgow Coma Scale but that uses a different concept in evaluating infants. Unlike different versions of the Glasgow Coma Scale, we include objective parameters such as the presence of lateralizing signs, pupillary abnormalities, and scalp injuries, all of which are easy to define. Being, in our opinion, more accurate in evaluating infants, this scale may help in the early diagnosis of intracranial disorders in apparently neurologically intact infants and may improve the estimation of prognosis in infants with apparently low CCS. We first presented the Trauma Infant Neurologic Score (TINS) at the International Neurotrauma Symposium in 1997 (Table ). In our opinion, TINS should include: (1) Mechanism of trauma (T); (2) whether or not the infant is intubated (I), because intubation makes proper neurologic assessment difficult; (3) three neurological (N) parameters (alertness vs. coma, lateralizing signs, and pupillary abnormalities); and (4) scalp injuries (S). The TINS suggested is simple to apply, short, and clear, scaling from 1 to 10 points. For each "bad" parameter, the infant earns one point. Because TINS is applied for trauma cases, the minimal score is 1 point (for minor trauma) (see Table 3). For severe mechanism of trauma (2 points), we include falls from more than 1 m, penetrating injuries, motor vehicle crashes, and severe blow injuries to the head. The maximal TINS, which is the worst possible, would be 10. Based on our preliminary experience from unpublished data , we assume that TINS < 4 is predictive of a good prognosis, TINS of 4 to 7 indicates moderate disability, and TINS > 8 would suggest poor prognosis. As for guidelines for CT in an infant with trauma, TINS of 2 or more would be the indication, in our opinion for CT. Of course, for patients at high risk (infants with hematologic or oncologic diseases), CT is performed in all cases. We think that TINS is more than another Glasgow Coma Scale score for children, because it emphasizes the unique aspect of clinical presentation and vulnerability of infants.

The usefulness and reliability of the suggested TINS is still to be determined in prospective studies of infants with head trauma and intracranial injuries. Using a different concept in building this score for infants, however, we hope to provide a better clinical and prognostic tool for this particular population.

ELIGIBILITY:
Inclusion Criteria:

* Age from birth till 24 months
* After Head Trauma (any type or severity)
* Arrival to Emergency room

Exclusion Criteria:

* None

Ages: 24 Hours to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants younger that 24 months who sustained head injury (Head Trauma)
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-04; Primary Completion 2018-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Neurological outcome at Discharge or within 1 month | up to 1 month
  clinical follow up and examination at discharge and clinics within 1 month after trauma

SECONDARY OUTCOMES:
Neurological outcome at 1 year after head injury in the Infant | up to 1 year after trauma
  clinical (and if available radiological follow up) 1 year after trauma

CONTACTS AND LOCATIONS:
Locations (1):
- Sharon Nechama, Laniado Hospital, Netanya, Israel, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hahn YS, Chyung C, Barthel MJ, Bailes J, Flannery AM, McLone DG. Head injuries in children under 36 months of age. Demography and outcome. Childs Nerv Syst. 1988 Feb;4(1):34-40. doi: 10.1007/BF00274081. PMID 3401866
- [Background] Raimondi AJ, Hirschauer J. Head injury in the infant and toddler. Coma scoring and outcome scale. Childs Brain. 1984;11(1):12-35. doi: 10.1159/000120157. PMID 6705608
- [Background] Morray JP, Tyler DC, Jones TK, Stuntz JT, Lemire RJ. Coma scale for use in brain-injured children. Crit Care Med. 1984 Dec;12(12):1018-20. doi: 10.1097/00003246-198412000-00002. PMID 6509997
- [Background] Reilly PL, Simpson DA, Sprod R, Thomas L. Assessing the conscious level in infants and young children: a paediatric version of the Glasgow Coma Scale. Childs Nerv Syst. 1988 Feb;4(1):30-3. doi: 10.1007/BF00274080. PMID 3135935
- [Background] Seshia SS, Seshia MM, Sachdeva RK. Coma in childhood. Dev Med Child Neurol. 1977 Oct;19(5):614-28. doi: 10.1111/j.1469-8749.1977.tb07995.x. No abstract available. PMID 913902
- [Background] Beni-Adani L, Flores I, Spektor S, Umansky F, Constantini S. Epidural hematoma in infants: a different entity? J Trauma. 1999 Feb;46(2):306-11. doi: 10.1097/00005373-199902000-00018. PMID 10029038
- [Background] Yi W, Liu R, Chen J, Tao S, Humphrey O, Bergenheim AT. Trauma infant neurologic score predicts the outcome of traumatic brain injury in infants. Pediatr Neurosurg. 2010;46(4):259-66. doi: 10.1159/000321800. Epub 2010 Dec 16. PMID 21160234